CLINICAL TRIAL: NCT07393542
Title: An Open Label, Randomized, Multicenter, Phase III Study of SHR-A2102 in Combination With Adebrelimab Versus Gemcitabine in Combination With Cisplatin/Carboplatin in Previously Untreated Locally Advanced or Metastatic Urothelial Carcinoma (NEC-UC2)
Brief Title: A Trial of SHR-A2102 With Adebrelimab in Locally Advanced or Metastatic Urothelial Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-302
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced or Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group 1 (Experimental): SHR-A2102 and Adebrelimab
  Interventions: Drug: SHR-A2102 and Adebrelimab
- Treatment group 2 (Experimental): SHR-A2102 and Adebrelimab
  Interventions: Drug: SHR-A2102 and Adebrelimab
- Treatment group 3 (Active Comparator): Gemcitabine and cisplatin / carboplatin
  Interventions: Drug: Gemcitabine and cisplatin / carboplatin

INTERVENTIONS:
Drug: SHR-A2102 and Adebrelimab — SHR-A2102 and Adebrelimab injection
  Arms: Treatment group 1; Treatment group 2
Drug: Gemcitabine and cisplatin / carboplatin — Gemcitabine injection and cisplatin injection / carboplatin injection
  Arms: Treatment group 3

SUMMARY:
The study is being conducted to evaluate the efficacy of SHR-A2102 with adebrelimab versus gemcitabine in combination with cisplatin/carboplatin in previously untreated locally advanced or metastatic urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to sign the informed consent form in writing.
2. Female or male, 18 to 80 years of age (both inclusive).
3. ECOG performance status of 0 or 1.
4. Expected survival of≥ 3 months.
5. Histologically confirmed diagnosis of urothelial carcinoma with radiographic or other confirmation of locally advanced unresectable or metastatic disease.
6. No prior systemic therapy for locally advanced or metastatic disease.
7. Able to provide archived or fresh tumor tissue for Nectin-4 and PD-L1 expression.
8. According to RECIST v1.1, there must be at least one measurable lesion;
9. Tolerant to cisplatin or carboplatin.
10. Adequate organ functions.
11. Agree to use medically approved contraceptive measures.

Exclusion Criteria:

1. Planned to receive any other anti-tumor therapy during the study.
2. Received other investigational products or treatments not yet marketed within 4 weeks.
3. Have received systemic anti-tumor treatment within 4 weeks;have received prior anti-tumor Chinese patent medicine treatment within 2 weeks; palliative radiotherapy or local therapy within 2 weeks.
4. Previously received therapy with an antibody-drug conjugate that meets any one of the following characteristics: targeting Nectin-4; containing irinotecan or its derivatives and acting as a topoisomerase I inhibitor.
5. Prior treatment with immune checkpoint inhibitors.
6. Major surgical procedure other than diagnostic or biopsy within 4 weeks, requiring elective surgery during the trial.
7. Active autoimmune disease requiring systemic treatment within 2 years.
8. Have experienced adverse events caused by previous anti-tumor treatments that have not recovered to grade ≤1 as per NCI-CTCAE v5.0.
9. Uncontrolled central nervous system metastases or carcinomatous meningitis.
10. Subjects with clinical symptoms or serous cavity effusion requiring puncture drainage.
11. Other malignancies within 5 years.
12. History of clinically significant pulmonary disease or any such disease suggested by chest imaging at screening.
13. Serious infections requiring intravenous antibiotics, antivirals, or antifungals for control.
14. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
15. History of immunodeficiency, or history of organ transplant.
16. Have experienced arteriovenous thrombosis or cardiovascular and cerebrovascular accidents within 6 months.
17. Subjects with clinically significant hemorrhage within 3 months.
18. Glycosylated hemoglobin (HbA1c) ≥ 8%.
19. Have serious cardiovascular and cerebrovascular diseases.
20. Allergic reaction to any component of the study treatment.
21. Subjects with active pulmonary tuberculosis.
22. Have severe dry eye, active keratitis, or corneal ulcer, or other conditions.
23. Female Subjects who are pregnant or planning to become pregnant during the study.
24. Other conditions unsuitable into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS), assessed by BICR | up to 50 months

SECONDARY OUTCOMES:
Determine the dose of SHR-A2102 in the second phase, participants included in the dose selection analysis were followed up at 6 months in the last case | Determine the dose of SHR-A2102 in the second phase, participants included in the dose selection analysis were followed up at 6 months in the last case
Overall Survival(OS) | up to 50 months
Objective response rate(ORR), assessed by BICR | up to 50 months
Disease control rate(DCR), assessed by BICR | up to 50 months
Duration of response(DoR), assessed by BICR | up to 50 months
PFS, assessed by investigator | up to 50 months
ORR, assessed by investigator | up to 50 months
DCR, assessed by investigator | up to 50 months
DoR, assessed by investigator | up to 50 months
Adverse event(AE) | up to 50 months
serious adverse event(SAE) | up to 50 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing C, China

IPD SHARING:
Plan to Share IPD: Undecided